CLINICAL TRIAL: NCT02559063
Title: Neurophysiological Aspects of Vision-based Speed of Processing Cognitive Training in Older Adults With Mild Cognitive Impairment
Brief Title: Vision-based Speed of Processing Cognitive Training and Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Vankee Lin, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1R01NR015452 (NIH); 1R01NR015452 (NIH)
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Mild Cognitive Impairment
Keywords: cognitive training; speed of processing; neuroplasticity; cognitive aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vision-based speed of processing (Experimental): Vision-based speed of processing training will use the INSIGHT online program (Posit Science), which includes five games (i.e., Eye for detail, Peripheral challenge, Visual sweep, Double decision, Target tracker) that practice processing speed and attention. All games share visual components, and the tasks become increasingly more difficult and require faster reaction times. Participants respond either by identifying what object they see or where they see it on the screen. The training will automatically adjust the difficulty of each task based on the participant's performance, ensuring that the participants always operate near their optimal capacity. The training programs will automatically record the percentage of completion of each game and scores.
  Interventions: Behavioral: Vision-based speed of processing training
- Mental leisure activities (Active Comparator): Mental leisure activities control activities were chosen to: 1) control for computer, online experience [and amount of time]; 2) not induce acute stress (i.e., without time management, speed component, or novel cognitive stimuli); 3) simulate participants' everyday mental activities; and 4) entertain participants to keep them from dropping out. Cross-word, Sudoku, and solitaire games will be used, which were also used in previous VSOP training study as control exercises. Participants can choose to practice any combination of games. At the end of their participation, the MLA control group will be provided with free 6-week access to the VSOP training program.
  Interventions: Behavioral: Mental leisure activities

INTERVENTIONS:
Behavioral: Vision-based speed of processing training — computerized cognitive tasks addressing vision-based speed of processing
  Arms: Vision-based speed of processing
Behavioral: Mental leisure activities — computerized cognitive tasks addressing different aspects of executive function
  Arms: Mental leisure activities

SUMMARY:
This project seeks to identify neural changes that occur in adults with mild cognitive impairment (MCI) after engagement in computerized cognitive training. In addition, this project aims to identify physiological factors that may bolster effects of the training on cognitive function. Individuals with MCI are at high risk for Alzheimer's disease (AD). Understanding how cognitive training protects cognitive function in MCI can contribute to development of effective interventions to slow progression to AD in individuals at risk, thereby reducing the significant morbidity and health care costs associated with AD.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI), especially amnestic type, is considered a symptomatic pre-Alzheimer's disease (AD) phase, and is prevalent in the aging population. Vision-based speed of processing (VSOP) cognitive training is one of the most widely applied behavioral interventions in community-dwelling older Americans free of AD, holding potential to slow cognitive decline. Its particular relevance to MCI is supported by converging evidence from our preliminary studies, including a recently completed pilot intervention study. However, we know little about the mechanisms underlying the benefits of VSOP training, limiting our ability to further exploit VSOP or other forms of cognitive training. In particular, we do not know if and how the effects of VSOP training on cognitive performance are mediated by neuroplasticity-related brain changes. Since recent evidence suggests that neuroplasticity is inducible throughout adult life, even in MCI, it is possible that VSOP training promotes neuroplasticity and slows neurodegeneration. In this early stage and new investigator application, we will focus on assessing whether and how VSOP training, relative to mental leisure activities (MLA), alters cognitive and neural functions in older adults with MCI, up to 6 months after training. The study will enroll and randomize 84 participants with amnestic MCI to VSOP training or MLA control groups. Three specific research aims are to (1) determine whether VSOP training improves processing speed and attention that are associated with changes of brain structural and functional connectivity; (2) test a novel neurophysiological pathway of VSOP training effect on brain structure and function; (3) examine the effect of VSOP training on untrained cognitive and functional domains and the role of neurophysiological changes underlying possible transfer effects. By examining multiple neural and novel physiological mechanisms linking a promising VSOP training intervention to improvements in cognitive performance, this application seeks to challenge and shift current research on cognitive training that merely examines training effects on cognitive outcomes. Discovery of neural, and physiological-related mechanisms in VSOP training will have important implications beyond this particular intervention. Findings from recent behavioral studies (e.g., cognitive intervention, physical exercise, nutrition, and bio-feedback intervention) suggest that for cognitive decline to be mitigated in individuals at risk for AD, it will be necessary for interventions to target the neural and peripheral physiological pathways that are susceptible to AD neuropathology. Confirmation of the study hypotheses could support immediate translation to clinical practices by demonstrating the efficacy, sustainability, and generalizability of cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of "mild cognitive impairment due to Alzheimer's disease" using the most recent NIA and Alzheimer's Association workshop criteria within 3 months: a) must have memory deficit (1-1.5SD below age- and education-corrected population norms); b) may have deficits in other cognitive domains (e.g., executive function); c) preserved BADL, defined as requiring occasional assistance on less than two items on the Minimum Data Set-Home Care interview, d) absence of dementia using NINCDS-ADRDA criteria;
* if on AD medication (i.e., memantine or cholinesterase inhibitors), no changes of doses in the 3 months prior to recruitment;
* capacity to give consent based on clinician assessment; and
* other: age ≥60 years, English-speaking, adequate visual acuity for testing, and community-dwelling.

Exclusion Criteria:

* current enrollment in another cognitive improvement study;
* major depression: 15-item Geriatric Depression Scale scored > 7;
* MRI contraindications, e.g., metallic implant, pacemaker, claustrophobia; and
* major vascular diseases: stroke, myocardial infarction, congestive heart failure.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Attention and processing speed test (UFOV) | change from baseline to 6-month follow-up

SECONDARY OUTCOMES:
Cognitive control and working memory (EXAMINER) | change from baseline to 6-month follow-up
instrumental activities of daily living (TIADL) | change from baseline to 6-month follow-up
mean of functional connectivity in default mode network | change from baseline to 6-month follow-up
  Resting state fMRI will be used to assess the functional connectivity of the neural network. SPM will be used to analyze and determine the change of the connectivity over time.
mean of structural connectivity in default mode network | change from baseline to 6-month follow-up
  Diffusion tensor imaging will be used to assess the structural connectivity of the neural network. FSL will be used to analyze and determine the change of the connectivity over time.

OTHER OUTCOMES:
long-term visual memory | change from baseline to 6-month follow-up
  long-term visual memory will be assessed using Brief Visuospatial Memory Test (BVMT)-R.

CONTACTS AND LOCATIONS:
Overall Officials: Vankee Lin, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Memory Care Program, Rochester, New York, United States